CLINICAL TRIAL: NCT05805384
Title: Evaluating a Noise Reduction Algorithm With Cochlear Implant Users
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-00815; SB1DC018761 (NIH)
Record Dates: First submitted 2023-03-23; First posted 2023-04-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hearing Impairment
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cochlear Implant Users (Experimental): Participants will complete up to 4 experiments evaluating the use of the Speech Enhancement using Dynamic thresholding Approach (SEDA) algorithm. Each testing session will take between 4-6 hours to complete. Testing sessions will continue until the completion of the experiments.
  Interventions: Device: SEDA

INTERVENTIONS:
Device: SEDA — Speech Enhancement using Dynamic thresholding Approach (SEDA) is a software algorithm that removes background noise.

SUMMARY:
In this study, a noise reduction algorithm will be implemented in various listening situations to evaluate its effectiveness in improving speech understanding for cochlear implant users ages 12 and older.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years of age.
* Be post-lingually deafened cochlear implant recipients with at least 6 months experience regardless of manufacturer.
* The PI must also deem the child to be developmentally able to complete the experiments.

Exclusion Criteria:

• Anyone who is not a cochlear implant user or is aged under 12 years.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Percent of Words Correctly Recognized in Noisy Conditions with SEDA NR | Up to Year 2 (Completion of Experiment 1.1)
  Participants will listen to sentences and repeat all the words they heard. This outcome measures the percent of words correctly recognized in noisy listening conditions while using the SEDA Noise Reduction (NR) algorithm.
Percent of Words Correctly Recognized in Noisy Conditions without NR | Up to Year 2 (Completion of Experiment 1.1)
  Participants will listen to sentences and repeat all the words they heard. This outcome measures the percent of words correctly recognized in noisy listening conditions without SEDA NR.
Percent of Words Correctly Recognized in Quiet Conditions with SEDA NR | Up to Year 2 (Completion of Experiment 1.1)
  Participants will listen to sentences and repeat all the words they heard. This outcome measures the percent of words correctly recognized in quiet listening conditions while using the SEDA NR.
Percent of Words Correctly Recognized in Quiet Conditions without NR | Up to Year 2 (Completion of Experiment 1.1)
  Participants will listen to sentences and repeat all the words they heard. This outcome measures the percent of words correctly recognized in quiet listening conditions with SEDA NR.
Visual Analogue Scale (VAS) Rating of SEDA NR | Up to Year 2 (Completion of Experiment 1.2)
  Participants will be presented with two buttons: one button will play a sample with SEDA NR and the other will play a sample without SEDA NR. Listeners will report which sample was preferable by clicking on a horizontal visual analog scale (VAS). VAS ratings will be scored on a scale of -10 to 10 where positive numbers indicate a preference for SEDA NR and negative numbers indicate a preference for not using SEDA NR. The magnitude of the absolute value of the score indicates the strength of the preference.
Percent of Words Correctly Recognized in Noisy Conditions with Clinical NR | Up to Year 2 (Completion of Experiment 2)
  Participants will listen to sentences and repeat all the words they heard. This outcome measures the percent of words correctly recognized in noisy listening conditions while using a clinical NR algorithm.
Percent of Words Correctly Recognized in Quiet Conditions with Clinical NR | Up to Year 2 (Completion of Experiment 2)
  Participants will listen to sentences and repeat all the words they heard. This outcome measures the percent of words correctly recognized in quite listening conditions while using a clinical NR algorithm.
Percent of Words Correctly Recognized with no SEDA NR | Up to Year 2 (Completion of Experiment 4)
  Participants will listen to sentences and repeat all the words they heard. This outcome measures the percent of words correctly recognized without SEDA NR.
Percent of Words Correctly Recognized with Standard SEDA NR | Up to Year 2 (Completion of Experiment 4)
  Participants will listen to sentences and repeat all the words they heard. This outcome measures the percent of words correctly recognized with Standard SEDA NR.
Percent of Words Correctly Recognized with Low-Computation SEDA NR | Up to Year 2 (Completion of Experiment 4)
  Participants will listen to sentences and repeat all the words they heard. This outcome measures the percent of words correctly recognized with the Low-Computation SEDA NR, which is designed to have minimal computation while maintaining an Extended Short-Time Objective Intelligibility Predictor (ESTOI) value similar to the "standard" SEDA implementation
Percent of Words Correctly Recognized with Very Low-Computation SEDA NR | Up to Year 2 (Completion of Experiment 4)
  Participants will listen to sentences and repeat all the words they heard. This outcome measures the percent of words correctly recognized with the Very Low-Computation SEDA NR, which is designed to have a reasonable ESTOI value with minimal computational requirements.

CONTACTS AND LOCATIONS:
Overall Officials: David M. Landsberger, Principal Investigator — NYU Langone Health
Locations (1):
- Tisch Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: David.landsberger@nyulangone.com. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to David.landsberger@nyulangone.com. To gain access, data requestors will need to sign a data access agreement.